CLINICAL TRIAL: NCT05824741
Title: Promoting Cardiovascular Health of Northern Appalachian Mother-Infant Dyads: PSU Infant Pilot Study
Brief Title: Early Intervention to Promote Cardiovascular Health of Mothers and Children (ENRICH)
Acronym: ENRICH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Ian M. Paul, M.D., M.Sc., Professor of Pediatrics and Public Health Sciences; Chief, Division of Academic General Pediatrics; Vice Chair of Faculty Affairs, Department of Pediatrics, Penn State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00021585; 1UG3HL162971-01 (NIH)
Record Dates: First submitted 2023-03-24; First posted 2023-04-24 (Actual); Results first posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Diseases; Infant ALL; Maternal Behavior; Childhood Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: This pilot study is being conducted to inform feasibility of the next phase of this research project.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): All participants will be enrolled into the intervention arm of this pilot study.
  Interventions: Behavioral: Infant Cardiovascular Health (CVH) Promotion

INTERVENTIONS:
Behavioral: Infant Cardiovascular Health (CVH) Promotion — The pilot infant CVH intervention will be delivered by Nurse-Family Partnership (NFP) staff starting no later than 1 month postpartum and lasting up to 6 months postpartum. The visit schedule will be consistent with the NFP visit structure to deliver intervention content at regularly scheduled visits that are typically 60 minutes long. This pilot study will include an enhanced version of the NFP standard care plan delivered by trained nurses to promote cardiovascular health by targeting soothing, feeding, sleep, and physical activity behaviors during infancy. The intervention delivered by trained visiting nurses will include behavior change strategies (e.g., goal setting, problem solving barriers). This pilot study will also examine the feasibility and acceptability of a digital device (infant foot worn actigraphy) during this same time period.

SUMMARY:
This pilot study aims to examine the feasibility and acceptability of adding a cardiovascular health module to the existing Nurse Family Partnership (NFP) home visitation program delivered by trained nurses in the Northern Appalachian region of Central Pennsylvania.

DETAILED DESCRIPTION:
The Promoting Cardiovascular Health of Northern Appalachian Mother-Infant Dyads: Pilot Study is a single arm pilot study that will enroll women with infants (<1 month of age) participating in the NFP home visitation program in the Northern Appalachian region of Central Pennsylvania. This pilot study will include an enhanced version of the NFP standard care plan delivered by trained nurses to promote cardiovascular health by targeting soothing, feeding, sleep, and physical activity behaviors during infancy. The intervention delivered by trained visiting nurses will include behavior change strategies (e.g., goal setting, problem solving barriers). This pilot study will also examine the feasibility and acceptability of a digital device (actigraphy) during this same time period.

ELIGIBILITY:
Inclusion Criteria:

1. Mother-infant dyad enrolled in and receiving the Nurse Family Partnership program through one of the study teams community partner offices throughout Central Pennsylvania
2. Mother age ≥ 18 years at time of delivery
3. Mother English speaking
4. Singleton infant born at ≥ 35 weeks' gestation
5. Infant age < 1 month at time of consent
6. Mother with reliable access to the internet for consent and data collection purposes

Exclusion Criteria:

1. Unable or unwilling to comply with the study visits and procedures.
2. Participation in a concurrent intervention study.
3. Infants with known chromosomal abnormalities, complex congenital heart disease, or birth defects inconsistent with survival to age 2 years.
4. Infant with substantial feeding difficulty (e.g., those requiring tube feeding)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian M Paul, MD, MSc, Principal Investigator — Penn State University
Locations (2):
- United States (2):
  - UPMC Home Health, Altoona, Pennsylvania
  - Geisinger, Danville, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Infants: All infants will be enrolled into the intervention arm of this pilot study.
  Infant Cardiovascular Health (CVH) Promotion: The pilot infant CVH intervention will be delivered by Nurse-Family Partnership (NFP) staff starting no later than 1 month postpartum and lasting up to 6 months postpartum. The visit schedule will be consistent with the NFP visit structure to deliver intervention content at regularly scheduled visits that are typically 60 minutes long. This pilot study will include an enhanced version of the NFP standard care plan delivered by trained nurses to promote cardiovascular health by targeting soothing, feeding, sleep, and physical activity behaviors during infancy. The intervention delivered by trained visiting nurses will include behavior change strategies (e.g., goal setting, problem solving barriers). This pilot study will also examine the feasibility and acceptability of a digital device (infant foot worn actigraphy) during this same time period.
Period: Overall Study
Arm/Group | Intervention Infants
Started | 15 (Number of infants)
Completed | 14 (Number of infants)
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group Infants: Behavioral intervention for parents of infants
Arm/Group | Intervention Group Infants
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants] — Population: Baseline data not collected on 1 participant
  Participants
    number analyzed (Participants) | 14
    <=18 years | 14
    Between 18 and 65 years | 0
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline data not collected on 1 participant so no information on race/ethnicity/sex
  Participants
    number analyzed (Participants) | 14
    Female | 10
    Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 4
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Integration of a Cardiovascular Health Module Into the Existing Nurse-Family Partnership (NFP) Home Visiting Program.
Description: Feasibility will be determined by acceptability of the curriculum to NFP nurses and participants as measured qualitatively through group discussion. Nurses will qualitatively provide feedback to the study team on whether they are able to successfully deliver new materials to their home visitation clients.
Time Frame: 6 months
Measure: Number; unit: participants receiving intervention
Arm/Group | Intervention
Number analyzed (Participants) | 14
participants receiving intervention | 14

2. Secondary Outcome: Number of Mothers Consenting for Their Infants to Participate in the Pilot Study.
Description: Enrollment feasibility will be determined by successful consent of 20 participants.
Time Frame: 6 months
Population: Participants enrolled
Measure: Number; unit: Participants enrolled
Arm/Group | Intervention Infants
Number analyzed (Participants) | 15
Participants enrolled | 15

3. Secondary Outcome: Utility of Infant Foot Worn Actigraphy Device for Infant Sleep Data Collection.
Description: Utility of device as demonstrated by days with complete sleep data.
Time Frame: 1 year
Reporting Status: Not Posted

4. Secondary Outcome: Number of Participants Completing Maternal Feeding Data Collection
Description: Determined by completion of study surveys.
Time Frame: 1 year
Reporting Status: Not Posted

5. Secondary Outcome: Participant Intervention Acceptability.
Description: Determined by completion of study qualitative surveys.
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Description: Infant adverse events
Groups:
- Intervention Group: Behavioral intervention for parents of infants
Arm/Group | Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-06-08): https://cdn.clinicaltrials.gov/large-docs/41/NCT05824741/Prot_SAP_ICF_000.pdf